CLINICAL TRIAL: NCT05376397
Title: Addressing Intersectional Stigma: Testing THRIVE 365 for Black Sexual Minority Men (On The Daily)
Brief Title: Testing THRIVE 365 for Black Sexual Minority Men (On The Daily)
Acronym: OTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Thrive Social Services (Other); Positive Impact Health Centers (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Devin English, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001082; K01MH118091 (NIH)
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Medication Adherence; Depressive Symptoms; Anxiety Symptoms; Emotion Regulation
MeSH Terms: conditions — Medication Adherence; Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iTHRIVE 365 (Experimental)
  Interventions: Behavioral: iTHRIVE 365

INTERVENTIONS:
Behavioral: iTHRIVE 365 — iTHRIVE 365 is a multicomponent intervention that combines mHealth features and institutional to support community priorities identified in formative CBPR. In line with best-practices for trials of intervention principles (TIPs) of interventions with mHealth features, THRIVE 365 deploys intervention elements that serve to accomplish intervention strategies. THRIVE 365 intervention strategies are to promote: 1)Health knowledge and motivation; 2)Social support coping; 3)Access to culturally-affirming healthcare; and 4)Housing and other economic resources. THRIVE 365 pursues these strategies via these intervention elements: 1)Weekly HIV and psychological health information and motivation content and daily health notifications; 2)Online moderated forums, interpersonal chats, and community calendars; 3)Linkage to biopsychosocial healthcare via THRIVE SS's network of BSMM-affirming providers; and 4)Housing and economic resources through THRIVE SS's direct support and referral network.

SUMMARY:
The primary goal of this study is to test a minority stress model of psychological health outcomes for Black sexual minority men (BSMM) while using and not using a novel intervention named THRIVE 365. THRIVE 365 combines mHealth and institutional support elements to provide four areas of support for BSMM: 1) Promote HIV and psychological health knowledge and motivation; 2) Foster a sense of community and positive social connections among BSMM; 3) Connect clients to BSMM-affirming healthcare, including HIV treatment and mental healthcare; 4) Provide resources for housing, transportation, and other economic empowerment. To examine the effects of the intervention, we will utilize a 14-day daily diary study to capture daily intervention engagement, HIV and psychological health outcomes, coping, and experiences of racial and sexual minority stressors. We will first examine main associations between intervention engagement and HIV (antiretroviral treatment use) and psychological health (depressive symptoms, anxiety symptoms, emotion regulation difficulties outcomes) outcomes, then consider how intervention engagement affects coping and attenuates the impacts of racial and sexual minority stressors during the 14 day period.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old or older ;
* Identifying as masculine
* Identifying as Black/African American
* Reporting being attracted to and/or sexually active with men;
* Able to complete all procedures in English.
* Mobile access to the internet in order to complete the once-daily survey procedures.

Exclusion Criteria:

* evidence of unstable, unmanaged, or serious psychiatric symptoms that could be made worse by participation;
* evidence of gross cognitive impairment that would interfere with successful completion of study procedures.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin English, PhD, Principal Investigator — Rutgers School of Public Health
Locations (1):
- Devin English, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that underlie the results reported in the article after deindentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following study publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] English D, Smith JC, Scott-Walker L, Lopez FG, Morris M, Reid M, Lashay C, Bridges D, McNeish D. Feasibility, Acceptability, and Preliminary HIV Care and Psychological Health Effects of iTHRIVE 365 for Black Same Gender Loving Men. J Acquir Immune Defic Syndr. 2023 May 1;93(1):55-63. doi: 10.1097/QAI.0000000000003167. PMID 36706362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iTHRIVE 365
Started | 34
Completed | 33
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Inclusion Criteria:
  16 years old or older ; Identifying as masculine Reporting being attracted to and/or sexually active with men; Able to complete all procedures in English. Mobile access to the internet in order to complete the once-daily survey procedures.
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 44 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 33
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Antiretroviral (ART) Medication Use
Description: A single dichotomous no(0)/yes(1) item assesses ART use over the past 24 hours: "In the past 24 hours, did you take ART medication?"
Time Frame: 24 Hours
Population: Men in the sample living with HIV
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 32
units on a scale | .94 (.24)

2. Primary Outcome: Depressive Symptoms
Description: The Patient Health Questionnaire-4 assesses anxiety and depressive symptoms. Participants rate the extent to which they had been experiencing each item the past day (e.g., "In the past 24 hours, I've been feeling down, depressed, or hopeless") on a scale from 0 (not at all) to 3 (completely). We used an average across all items for each time point.
Time Frame: 24 Hours
Population: All Participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 34
Score on a scale | .39 (.62)

3. Primary Outcome: Anxiety Symptoms
Description: The Patient Health Questionnaire-4 assesses anxiety and depressive symptoms. Participants rate the extent to which they had been experiencing each item the past day (e.g., "In the past 24 hours, I've been feeling nervous, anxious, or on edge") on a scale from 0 (not at all) to 3 (completely). We used an average across all items for each time point.
Time Frame: 24 Hours
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 34
units on a scale | .43 (.66)

4. Primary Outcome: Emotion Regulation
Description: A validated four-item version of the Difficulties with Emotion Regulation Scale assesses emotion regulation. Participants rated the extent to which they had been experiencing each item (e.g., "In the past 24 hours, I've been experiencing my emotions as overwhelming") in the past day on a scale from 0 (not at all) to 3 (completely). We used an average across all items for each time point.
Time Frame: 24 Hours
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 34
units on a scale | .48 (.51)

5. Secondary Outcome: Coping
Description: A modified version of the Brief-COPE assesses coping approaches to stress over the last 24 hour. It includes the 3 items from the interconnectedness and 3 items problem-oriented subscales (Greer, 2007), and 3 original items assessing specific interconnectedness with Black LGBTQ people and problem-oriented action against injustice ("I've connected with another Black LGBTQ person for support", "I've spoken out against negative treatment", "I've posted about injustice on social media"). Participant indicate all the coping approaches among the 9 total that they utilized over the last 24 hours (Range: 0-9 coping approaches).
Time Frame: 24 Hours
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iTHRIVE 365
Number analyzed (Participants) | 34
units on a scale | 2.14 (1.83)

ADVERSE EVENTS:
Time Frame: Two weeks
Description: This was classified as minimal risk in IRB review. As such, there were no participants at-risk for serious adverse events, all-cause mortality, or other adverse events.
Arm/Group | iTHRIVE 365
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT05376397/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT05376397/SAP_001.pdf